CLINICAL TRIAL: NCT05876039
Title: Comparison of Two Dosage of Remifentanil Infusion Combined with Propofol-based Total Intravenous Anesthesia in Percutaneous Vertebroplasty
Brief Title: Optimal Dosage of Remifentanil for Vertebroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Cheng Tseng, Principal Investigator, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 210705163-V3
Record Dates: First submitted 2023-05-03; First posted 2023-05-25 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2023-05

CONDITIONS: Remifentanil; Analgesia
Keywords: Vertebroplasty; Remifentanil; Target-controlled infusion; Procedural analgesia and sedation
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group remifentanil of 1.0 ng/mL (Experimental): Initial remifentanil effect-site concentration of 1.0 ng/mL
  Interventions: Drug: Initial remifentanil effect-site concentration
- Group remifentanil 2.0 ng/mL (Active Comparator): Initial remifentanil effect-site concentration of 2.0 ng/mL
  Interventions: Drug: Initial remifentanil effect-site concentration

INTERVENTIONS:
Drug: Initial remifentanil effect-site concentration — Different initial remifentanil effect-site concentration

SUMMARY:
Percutaneous vertebroplasty has become a mainstay in the management of osteoporotic and malignant vertebral fractures. Procedural analgesia and sedation (PAS) with propofol and remifentanil may provides optimal hypnotic and analgesic effects.

DETAILED DESCRIPTION:
Percutaneous vertebroplasty has become a mainstay in the management of osteoporotic and malignant vertebral fractures. Many anesthetic methods have been used in percutaneous vertebroplasty; however, there is no gold-standard method. Procedural analgesia and sedation (PAS) are one of the commonly used approaches. For its unique properties, including rapid onset, precise intraoperative control, and a fast recovery profile, remifentanil is preferable to other opioids administration in a target-controlled infusion (TCI) pump. Combination of remifentanil with propofol may improve sedation experience; however, it can increase a risk of respiratory depression. Moreover, propofol and remifentanil are often administered with 2 TCI pumps to, respectively, provide hypnotic and analgesic effects, which together are considered to be an ideal anesthetic technique.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score of I-III patients receiving percutaneous vertebroplasty under procedural sedation and analgesia with remifentanil and propofol

Exclusion Criteria:

* Age < 20 or > 80 years
* ASA classifications > III
* Pregnancy
* Known allergies to opioids, propofol or any drugs used in the study
* Emergency surgery
* Patient refusal

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Adequate analgesia at the time of the trocar needle insertion | Time at the trocar needle placement
  Remaining moveless at the time of the trocar needle insertion
Adequate analgesia at the time of the bone cement injection | Time at the bone cement injection
  Remaining moveless at the time of the bone cement injection

SECONDARY OUTCOMES:
Hypotension at the time of the trocar needle placement | Time at the trocar needle placement
  Mean blood pressure > 30% decrease from baseline
Hypotension at the time of the bone cement injection | Time at the bone cement injection
  Mean blood pressure > 30% decrease from baseline
Apnea with desaturation at the time of the trocar needle placement | Time at the trocar needle placement
  Oxygen saturation < 95%
Apnea with desaturation at the time of the bone cement injection | Time at the bone cement injection
  Oxygen saturation < 95%
TCI pump adjustments at the time of the trocar needle placement | Time at the trocar needle placement
  Frequency of TCI pump adjustments
TCI pump adjustments at the time of the bone cement injection | Time at the bone cement injection
  Frequency of TCI pump adjustments
Numeric rating scale | Postoperative one hour
  Postoperative numeric rating scale. NRS scores is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Lai HC, Chen CL, Huang YH, Wu KL, Huang RC, Lin BF, Chan SM, Wu ZF. Comparison of 2 effect-site concentrations of remifentanil with midazolam during transrectal ultrasound-guided prostate biopsy under procedural analgesia and sedation: A randomized controlled study. Medicine (Baltimore). 2022 Sep 9;101(36):e30466. doi: 10.1097/MD.0000000000030466. PMID 36086764
- [Background] Lai HC, Tsai YT, Huang YH, Wu KL, Huang RC, Lin BF, Chan SM, Wu ZF. Comparison of 2 effect-site concentrations of remifentanil with midazolam during percutaneous transluminal balloon angioplasty under monitored anesthesia care: A randomized controlled study. Medicine (Baltimore). 2021 Jul 30;100(30):e26780. doi: 10.1097/MD.0000000000026780. PMID 34397727
- [Background] Cannata F, Spinoglio A, Di Marco P, Luzi M, Canneti A, Ricciuti G, Reale C. Total intravenous anesthesia using remifentanil in extracorporeal shock wave lithotripsy (ESWL). Comparison of two dosages: a randomized clinical trial. Minerva Anestesiol. 2014 Jan;80(1):58-65. Epub 2013 Jul 9. PMID 23839319